CLINICAL TRIAL: NCT00364676
Title: A Phase 1 Study of Vinorelbine Liposomes Injection (VLI) for Treatment in Patients With Advanced Solid Tumors, Non-Hodgkin's Lymphoma or Hodgkin's Disease
Brief Title: Study of Vinorelbine Liposomes Injection for Advanced Solid Tumors, Non-Hodgkin's Lymphoma or Hodgkin's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS501
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Tumors; Hodgkins Disease; Non-Hodgkins Lymphoma
Keywords: Vinorelbine; solid tumors; Hodgkins; Non hodgkins; Lymphoma; Advanced solid tumors
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma

ARMS (2):
- 1 (Experimental): Patients are dosed on Day 1 and Day 8 of a 21-day cycle.
  Interventions: Drug: VLI
- 2 (Experimental): Patients are dosed on Day 1 of a 21-day cycle.
  Interventions: Drug: VLI

INTERVENTIONS:
Drug: VLI — Patients are dosed on Day 1 and Day 8 of a 21-day cycle.
  Arms: 1
Drug: VLI — Patients are dosed on Day 1 of a 21-day cycle.
  Arms: 2

SUMMARY:
This Phase 1 study will determine the safety, tolerability, and pharmacokinetics of vinorelbine liposomes injection (VLI) in patients with advanced solid tumors, non-Hodgkin's lymphoma, or Hodgkin's disease.

DETAILED DESCRIPTION:
The objectives of this study are:

* To assess the safety and tolerability of treatment with VLI.
* To determine the maximum tolerated dose (MTD) of VLI.
* To characterize the pharmacokinetic (PK) profile of VLI.
* To explore preliminary tumor response of VLI.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor refractory to standard therapy or for which no standard therapy is known to exist, or relapsed and/or refractory non-Hodgkin's lymphoma or Hodgkin's disease
2. Adequate hematologic, hepatic and renal functions as defined by laboratory tests.
3. At least 18 years of age.
4. Have a life expectancy of at least 12 weeks.
5. Patients must give written informed consent.
6. ECOG or Zubrod performance status of 0, 1, or 2.

Exclusion Criteria:

1. Primary tumors of central nervous system (CNS). Symptomatic brain metastases (unless patient is stable without requirement of steroids and/or antiseizure medications for at least 3 months) or leptomeningeal tumor involvement.
2. Prior chemotherapy or radiotherapy within 4 weeks prior to study entry (6 weeks for nitrosoureas and mitomycin C).
3. Planned concurrent systemic therapy and/or radiotherapy drug study treatment.
4. Use of investigational drugs, biologics or devices within 28 days prior to study treatment or planned use during the course of the study.
5. Active infection or any serious underlying medical condition, which would impair the ability of the patient to receive protocol treatment.
6. Prophylactic hematologic growth factors administered less than or equal to 2 weeks prior to start of therapy with VLI (excluding darbepoetin alfa, epoetin alfa).
7. Female patients who are pregnant or lactating.
8. Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-07; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of VLI. | 21 Days

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, MD, Principal Investigator — Cancer Therapy and Research Center, Texas; Gerald Batist, MD, Principal Investigator — McGill Centre for Translational Research in Cancer-Jewish General Hospital Clinical Research Unit; Anthony W. Tolcher, MD, Principal Investigator — South Texas Accelerated Research Therapeutics
Locations (3):
- United States (2):
  - Cancer Therapy and Research Center, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- McGill Centre for Translational Research in Cancer-Jewish General Hospital Clinical Research Unit, Montreal, Quebec, Canada